CLINICAL TRIAL: NCT05936723
Title: Influence of Different Methods of Respiratory Muscle Training on Athletic Performance and Pulmonary Function in Short-track Speedskaters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Institute of Sport - National Research Institute, Poland (Other)
Responsible Party: Principal Investigator, Tomasz Kowalski, Principal Investigator, Institute of Sport - National Research Institute, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TK01/2023
Record Dates: First submitted 2023-06-22; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Respiratory Muscle Training

STUDY DESIGN:
Intervention Model Description: parallel group-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voluntary Isocapnic Hyperpnoea (VIH) (Active Comparator): Group performing respiratory muscle training with Voluntary Isocapnic Hyperpnoea (VIH) method.
  Interventions: Behavioral: Respiratory Muscle Training - VIH
- Inspiratory Pressure Threshold Loading (IPTL) (Active Comparator): Group performing respiratory muscle training with Inspiratory Pressure Threshold Loading (IPTL) method.
  Interventions: Behavioral: Respiratory Muscle Training - ITPL

INTERVENTIONS:
Behavioral: Respiratory Muscle Training - VIH — The VIH group will train every second day with gradual progression based on session length and breathing frequency. Participants will begin with 3 minutes of exercise with a frequency of 20 breaths·min-1 during the first session and add no more than 1 minute or 2 breaths·min-1 with each consecutive session.
  Arms: Voluntary Isocapnic Hyperpnoea (VIH)
Behavioral: Respiratory Muscle Training - ITPL — The IPTL group will train 5 days a week, twice a day, with at least 6 hours break between sessions. The session will consist of 30 dynamic inspiratory maneuvers with progressive overload based on gradually increased resistance. The VIH group will train every second day with gradual progression based on session length and breathing frequency. Participants will begin with 3 minutes of exercise with a frequency of 20 breaths·min-1 during the first session and add no more than 1 minute or 2 breaths·min-1 with each consecutive session.
  Arms: Inspiratory Pressure Threshold Loading (IPTL)

SUMMARY:
This research aims to explore the impact of two distinct methods of respiratory muscle training, voluntary isocapnic hyperpnoea (VIH) and inspiratory pressure threshold loading (IPTL), on athletic performance and pulmonary function in short-track speedkaters. The study will employ a parallel group-randomized trial design and will span a period of six weeks, during which participants will undergo regular, partially supervised training sessions.

The primary objective of the research is to assess the changes in athletic performance resulting from respiratory muscle training using VIH and IPTL techniques. Athletic performance will be measured through a range of standardized performance tests relevant to the participants' specific sporting activities (Wingate Test, CPET, on-ice time-trial performance). Pulmonary function will be measured by spirometry examination.

The group will consist of healthy, highly-trained professional short-track speedskaters.

DETAILED DESCRIPTION:
This study aims to investigate the effects of two different respiratory muscle training methods, namely voluntary isocapnic hyperpnoea (VIH) and inspiratory pressure threshold loading (IPTL), on athletic performance and pulmonary function. The research will adopt a parallel group-randomized trial design, spanning a six-week period of regular, partially supervised training sessions.

The primary objective is to evaluate changes in athletic performance resulting from respiratory muscle training using VIH and IPTL techniques. Standardized performance tests relevant to the participants' specific sports will be utilized (Wingate Test, CPET, on-ice time-trial performance).

In addition, the impact of respiratory muscle training on pulmonary function will be assessed, focusing on parameters such as forced vital capacity (FVC), forced expiratory volume in one second (FEV1), peak expiratory flow (PEF). These measurements will provide insights into the potential enhancements of respiratory muscle strength and function through VIH and IPTL.

Participants will be randomly assigned to either the VIH or IPTL training group. Regular training sessions will be conducted under partial supervision to ensure proper technique and adherence. Close monitoring will be implemented to track progress and identify any potential adverse effects.

The findings of this research will hold implications for athletes and individuals seeking to optimize their athletic performance and respiratory muscle function. By comparing the effects of VIH and IPTL, the study aims to identify the most effective respiratory muscle training method.

Ultimately, this research will contribute to the existing knowledge on respiratory muscle training and its potential benefits for athletes and individuals engaged in physical activities. The results obtained will provide evidence-based guidance for the development of targeted training protocols that can enhance athletic performance and respiratory health.

ELIGIBILITY:
Inclusion Criteria:

* valid medical certificate to compete sports professionally,
* lack of ongoing medication intake,
* lack of any medical condition,
* lack of previous experience with RMT,
* performance caliber corresponding to at Elite/World Class (Participant Classification Framework, McKay 2022).

Exclusion Criteria:

* any ongoing medication intake or medical condition.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Maximum Power in Wingate Test | before and after the intervention (6-weeks)
  Difference between maximum power achieved in Wingate Test in Week 1 and maximum power achieved in Wingate Test in Week 6 of the intervention. Unit: watts per kg
Changes in Total Work in Wingate Test | before and after the intervention (6-weeks)
  Difference between total work performed in Wingate Test in Week 1 and total work performed in Wingate Test in Week 6 of the intervention. Unit: kilojouls
Changes in VO2max measured with cycloergometer cardiopulmonary exercise testing | before and after the intervention (6-weeks)
  Difference between VO2 measured in Week 1 and VO2 measured in Week 6 of the intervention. Unit: mL/min/kg.
Changes in forced volume vital capacity (FVC) measured with spirometry test | before and after the intervention (6-weeks)
  Difference between FVC measured in Week 1 and FVC measured in Week 6 of the intervention. Unit: litres.
Changes in on-ice performance measured with time trial effort | before and after the intervention (6-weeks)
  Changes in time achieved during on-ice time trial performance in Week 1 and time achieved during on-ice time trial performance in Week 6 of the intervention. Unit: time in seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sport - National Research Institute, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No